CLINICAL TRIAL: NCT03758469
Title: A Single-Center, Open-Label, Randomized, Two-Stage, Two-Way Crossover Study Evaluating Drug-Drug Interaction (DDI) Between HSK3486 Injectable Emulsion and Rifampin Capsules in Healthy Subjects.
Brief Title: A Study Evaluating Drug-Drug Interaction (DDI) Between HSK3486 Injectable Emulsion and Rifampin Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-103
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): 0.4 mg/kg
  Interventions: Drug: HSK3486
- rifampin , HSK3486 (Experimental): 600 mg;0.4 mg/kg
  Interventions: Drug: rifampin , HSK3486

INTERVENTIONS:
Drug: HSK3486 — Sequence 1: Intravenously infuse 0.4 mg/kg HSK3486 in the morning on an empty stomach. Complete infusion within 1 min.
  Arms: HSK3486
Drug: rifampin , HSK3486 — Sequence 2: Orally take 600 mg rifampin once a day for 8 consecutive days in the morning on an empty stomach, followed by 1 min intravenous infusion of 0.4 mg/kg HSK3486 30 min later.
  Arms: rifampin , HSK3486

SUMMARY:
This is a Phase I, single-center, open-label, randomized,two-way crossover, propofol-controlled, two-stage study evaluating the safety and pharmacokinetics/pharmacodynamics of IV maintenance dose and IV single loade dose plus maintenance dose of HSK3486 emulsion for injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females with full capacity for civil conduct, aged ≥18 and ≤45 years old. Both male and female subjects should be enrolled;
2. Male subjects weighing ≥50 kg, female subjects weighing ≥45 kg. All subjects should have a body mass index (BMI) of ≥19.0 and ≤26.0 kg/m2;
3. Blood pressure between 100-139/60-89 mmHg; heart rate between 60-99 beats/min; body temperature between 35.8-37.5 °C; respiratory rate between 12-20 breaths/min; SpO2 when inhaling ≥95%;
4. Normal physical examinations, laboratory examinations (blood routine, blood biochemistry and urine routine), and 12-lead electrocardiogram (ECG), or abnormal but without clinical significance as judged by the investigators; no significantly potential difficult airway (modified Mallampati score I-II);
5. No previous history of major organ primary diseases, such as liver, kidneys, digestive tract, blood, and metabolic diseases; no history of malignant hyperthermia and other genetic conditions; no history of mental/neurological diseases; no history of epilepsy; no contraindications for deep sedation/general anesthesia; no clinically significant history of anesthesia accidents;
6. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with trial protocol.

Exclusion Criteria:

1. Known sensitivity to excipients in HSK3486 injectable emulsion (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate and sodium hydroxide), rifampin, or contraindications mentioned in the prescribing information of rifampin; history of drug allergies (including anesthetics), allergic diseases, or those with hyperactive immune response;
2. In receipt of any one of the following medications or treatments during screening/baseline:

   1. History of drug abuse or any signs of chronic benzodiazepines use (such as insomnia, anxiety, spasms) within 3 months prior to screening, or a positive urine drug test during baseline;
   2. Participated in clinical trials involving any medications or medical devices within 3 months prior to screening, or subjects who have participated in 3 or more drug clinical trials within the past year;
   3. In receipt of rifampin within 4 weeks prior to screening;
   4. Serious infection, trauma or major surgery within 4 weeks prior to screening; or acute disease with clinical significance (determined by the investigator) within 2 weeks prior to screening, including GI diseases or infections (such as respiratory or CNS infections);
   5. In receipt of propofol, other sedatives/anesthetics and/or opioid analgesics or compounds containing analgesics within 1 week prior to baseline;
   6. In receipt of prescription drugs, Chinese herbal medicines, over-the-counter drugs or food supplements (such as vitamins and calcium supplements) other than contraceptives, paracetamol, oral non-steroidal anti-inflammatory drugs, topical over-the-counter preparations, within 2 weeks prior to baseline; unless the principal investigator (PI) and the sponsor agree that the medication has no effect on the safety and PK/PD results of the trial;
3. A history or evidence of any one of the following diseases prior to screening/baseline:

   1. History of cardiovascular diseases such as: postural hypotension, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, tachycardia/bradycardia requiring medication, third-degree atrioventricular block or QTcF interval ≥450 ms (Fridericia's correction formula);
   2. Respiratory insufficiency, history of obstructive pulmonary disease, history of asthma, sleep apnea; history of failed tracheal intubation; history of bronchospasm requiring treatment within 3 months prior to screening; acute respiratory infection, and with obvious symptoms such as fever, wheezing, nasal congestion or cough within 1 week prior to baseline;
   3. History of GI tract diseases: Gastrointestinal obstruction, active GI bleed, potential for reflux and aspiration;
4. Laboratory results that meet any of the following during screening/baseline:

   1. Positive result for either HBsAg, HCV, HIV, or syphilis;
   2. Abnormal hepatic or renal function confirmed after re-examination;

      * ALT or AST > 1×ULN;
      * Creatinine > 1×ULN;
      * TBIL > 1.0×ULN;
5. History of alcohol abuse within 3 months prior to screening, abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or positive result for breath alcohol test during baseline;
6. Smoke more than 5 cigarettes per day and a total of more than 60 cigarettes within 3 months prior to screening;
7. Blood donation or blood loss ≥200 mL within 30 days prior to screening; plasma donation or plasma exchange within 7 days prior to screening;
8. Subjects who consume any beverages or foods containing alcohol, grapefruit juice or methylxanthine (such as coffee, tea, coca-cola, chocolate, functional drinks), to participate in strenuous physical activities and other factors that may affect drug absorption, distribution, metabolism, and excretion within 2 days prior to enrollment; subjects who are unable to fast for 8 hours prior to dose administration;
9. Subjects expected to have surgery or hospitalization during the trial;
10. Subjects unsuitable for arterial blood collection, such as subjects who have positive Allen's test;
11. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial; subjects who are planning pregnancy within 1 month after the completion of the trial (including male subjects);
12. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | From the start of HSK3486 administration to 24 h after the start of administration on day 1
Area under the concentration-time curve (AUC0-t, AUC0-∞) | From the start of HSK3486 administration to 24 h after the start of administration on day 1

SECONDARY OUTCOMES:
Terminal elimination half life (t1/2) | From the start of HSK3486 administration to 24 h after the start of administration on day 1
Time to fully awake | From the start of HSK3486 administration until the subjects is fully awake on day 1
MOAA/S(modified observer's assessment of alert /sedation)-time curve | From the start of HSK3486 administration until the subjects is fully awake on day 1
  Observe the change of modified observer's assessment of alert /sedation during the whole trial
BIS(bispectral index)-time curve | From the start of HSK3486 administration to 60 min after the start of administration on day 1
  Observe the changes of bispectral index during the whole trial
Blood pressure | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of blood pressure during the whole trial
Heart rate | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of heart rate during the whole trial
Respiratory rate or blood oxygen saturation | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of respiratory rate or blood oxygen saturation during the whole trial
Blood routine test | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of blood routine test during the whole trial
Urine routine test | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of urine routine test during the whole trial
Blood biochemical examination | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of Blood biochemical examination during the whole trial
12-Electrocardiogram | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Observe the changes of heart rate, RR interval, QT interval , QTcF interval , PR interval and QRS interval of electrocardiogram during the whole trial
Number of patients with adverse events | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Safety endpoits
Concurrent medications | From the start of HSK3486 administration to 24 h after the start of administration on day 1
  Safety endpoits

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, China